CLINICAL TRIAL: NCT01688570
Title: Mechanisms of Neuromuscular Fatigue Post Stroke
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Phillip Nelson, MD, Assistant Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: UL1RR031973-02 (NIH)
Record Dates: First submitted 2012-09-12; First posted 2012-09-20 (Estimated); Last update posted 2015-11-05 (Estimated); Status verified 2015-11

CONDITIONS: Stroke
Keywords: neuromuscular fatigue; motor impairment
MeSH Terms: conditions — Stroke | interventions — Duloxetine Hydrochloride; Cyproheptadine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Duloxetine (Active Comparator): Neuromuscular fatigue testing with duloxetine dose
  Interventions: Drug: duloxetine
- Cyproheptadine (Active Comparator): Neuromuscular fatigue testing with cyproheptadine dose
  Interventions: Drug: Cyproheptadine
- Placebo (Placebo Comparator): Neuromuscular fatigue testing with placebo dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: duloxetine — Single dose, orally (pill), 30 mg, taken 6 hours prior to start of the testing session. Subjects will only take a single dose of duloxetine once.
  Other Names: Cymbalta
  Arms: Duloxetine
Drug: Cyproheptadine — Single dose, orally, 8 mg, 6 hours prior to the start of the respective testing session. Subjects will take a single dose of cyproheptadine once.
  Arms: Cyproheptadine
Drug: Placebo — Single dose, orally, 6 hours prior to the start of the respective testing session. Subjects take a single dose once.
  Arms: Placebo

SUMMARY:
While baseline weakness is clearly an important factor that contributes to disability post stroke, neuromuscular fatigue (the acute reduction in force production) of the paretic musculature likely compounds strength deficits and further exacerbates disability. The proposed study aims to improve our understanding of the mechanisms of neuromuscular fatigue in people post stroke in order to optimize strength training. In healthy individuals, both central (neural) and peripheral (muscle) factors are determinants of neuromuscular fatigue, but preliminary data from our laboratory suggests a greater contribution of central components to neuromuscular fatigue in the paretic musculature. Although cortical pathways are clearly disrupted post stroke, it is likely that brainstem pathways, known to have neuromodulatory effects on spinal motor circuitry, are more involved in the sustaining of force in the paretic leg, compared to the non-paretic and control legs. Therefore, the purpose of this proposal is to examine the role of descending neuromodulatory pathways of the brainstem in neuromuscular fatigue post stroke (Aim 1) and to correlate brainstem-related changes in neuromuscular fatigue to walking function (Aim 2). The investigators propose that stroke survivors' decreased capability to sustain force overtime results from the diminished ability of spinal motoneurons to respond to brainstem neuromodulatory inputs (serotonin (5-HT) and norepinephrine (NE)). Aim 1 will quantify stroke-related decreases in motor output sensitivity to a 5-HT and NE reuptake inhibitor (SNRI), serotonin antagonist, or placebo during sub-maximal intermittent fatiguing knee extension contractions. If motoneurons are desensitized to descending monoamines in chronic stroke patients, then they will be less sensitive to the effects of drugs that increase monoamine levels. The investigators predict that in response to the SNRI or serotonin antagonist, the paretic leg will show less change in time to task failure and a smaller reduction in strength as compared to the non-paretic and control legs. For Aim 2, the investigators predict that stroke subjects with the highest walking function will demonstrate the greatest fatigue-related changes in response to the SNRI. This proposal adopts an innovative model of motor impairment post stroke by including the role of subcortical structures in neuromuscular fatigue.

ELIGIBILITY:
Inclusion Criteria:

General

* be at least 18 years of age
* Cognitively able to give informed consent Stroke

  -≥ 6 months post diagnosis of unilateral cortical stroke
* residual leg paresis

Exclusion Criteria:

General

* chronic low back or hip pain
* major psychiatric disorders (e.g. depression
* substance abuse
* head trauma
* neurodegenerative disorder
* any uncontrolled medical disorder (e.g. hypertension)
* taking any medication or supplement (e.g. St. John's Wort) that has 5-HT or NE mechanisms of action(including Monoamine oxidase inhibitors (MAO) inhibitors)
* narrow angle glaucoma
* chronic liver or kidney disorders Stroke
* history of multiple strokes
* people who are unable to follow 2 step commands
* people who cannot walk ≥ 10 ft without physical assistance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2011-08; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Force generation | At time of each of 4 testing sessions (all sessions within a 2 year period).
  Sub-maximal and maximal force measurements will be made during brief contractions during each of the four testing sessions. All sessions will occur at least one week apart and within a total time span of 2 years.

SECONDARY OUTCOMES:
Surface electromyography (EMG)of lower leg muscles. | EMG measurements will be made during each of the four sessions.
  Sessions will occur at least a week apart and within a 2 year time span.

CONTACTS AND LOCATIONS:
Overall Officials: Philip A. Nelson, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States